## Train Your Brain: A Pilot Project to Improve Memory and Decision Making NCT05879198

Final Approved Protocol

Document Date 8/16/2024

## **Data Analytic Plan**

Primary Outcomes: Changes in delay discounting, time horizon, and executive functions.

Descriptive statistics will be used to characterize the sample and psychometric properties will be examined (reliability, etc.). Changes in quantitative measures (including delay discounting, time horizon, and executive functions) will be examined in a number of ways. First, we will examine each variable to evaluate mean, standard deviations, skew and kurtosis. We will examine the overall number of youth who demonstrated decreases in delay discounting (5-Trial Adjusting Measure of Delay Discounting). We will use t-tests and reliable change indices (RCI) to examine differences in mean levels of consideration of future consequences (Consideration of Future Consequences Scale) and measures of executive function (Tower of Hanoi, Letter Number Sequencing, Iowa Gambling Task). We will set statistical significance at p<.05.

Secondary Outcomes: Changes in risk behaviors.

Descriptive statistics will also be examined for all secondary outcomes. We will then evaluate changes in our measures of risky behaviors (the Youth Risk Behavior Survey and the Alcohol and Marijuana Expectancies measures) using t-tests and RCIs. We will set statistical significance at p<.05.